CLINICAL TRIAL: NCT05835960
Title: The Role of Early Diagnosis and Treatment of Anal Intraepithelial Neoplasia in the Prevention of Anal Squamous Cell Carcinoma: Identifying Prognostic Biomarkers.
Brief Title: Anal Intraepithelial Neoplasia and Anal Squamous Cell Carcinoma
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Imperial College London (Other)
Responsible Party: Sponsor
Other Study IDs: 234715
Record Dates: First submitted 2023-04-19; First posted 2023-04-28 (Actual); Last update posted 2023-04-28 (Actual); Status verified 2023-04

CONDITIONS: Anal Cancer; Anal Squamous Intraepithelial Neoplasia
Keywords: Anal Cancer; Early Diagnosis; Anal Squamous Intraepithelial Lesion; Biomarker; HPV; Treatment response
MeSH Terms: conditions — Anus Neoplasms; Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood samples, FFPE and frozen biopsies of anal high-grade squamous intraepithelial lesions, FFPE and frozen biopsies of anal squamous cell carcinoma, normal control tissue.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This is a study involving exome sequencing and immune profiling of matched tissue and blood samples from patients with both high-grade squamous intraepithelial lesions and anal squamous cell carcinoma. This is a collaborative project between Imperial College London and the Institute of Cancer Research (ICR), investigating the genetic predeterminants for the progression of anal HSIL to SCC as well as the immunogenetic profile of these conditions will be beneficial for risk stratification (with respect to identifying those individuals with anal HSIL most likely to progress to invasive disease), the identification of potential new drug targets and will add to our understanding of how the tumour microenvironment may influence treatment response and disease recurrence of both anal HSIL and SCC.

DETAILED DESCRIPTION:
Patients, as identified by the colorectal MDT, are approached, and consented for tissue and blood collection on the day of their diagnostic procedure; the plasma and buffy coat are extracted from the EDTA tubes. A tissue biopsy is performed adjacent to the area sampled for diagnosis and flash frozen in liquid nitrogen. Once the diagnosis of anal cancer is confirmed, the FFPE diagnostic tissue, is requested from the Tissue Bank for the study.

The FFPE and the fresh frozen tissue samples are sliced and put on slides. Stained slides are reviewed by a consultant histopathologist, areas of anal HSIL and SCC are marked.

All samples are transferred to the ICR. Tumour DNA and RNA are extracted from the tissue samples and germline DNA from the buffy coat of the blood sample.

Exome sequencing followed by Bioinformatic analysis is carried out where somatic mutations are evaluated for impact on gene expression and compared between germline, anal HSIL and SCC samples. After a quality control process is complete, the entire dataset is compared with the germline DNA reads, thereby identifying somatic mutations. Candidate mutations are finally cross-referenced with the Cancer Genome Census and string analysis of relevant mutations is performed to assess for cancerogenic impact.

Bulk RNA and targeted RNA based T-Cell Receptor (TCR) sequencing will be carried out, with TCR sequencing also being performed on the blood. This will establish which immune cell types are present in the SCC vs HSIL (by transcriptomic deconvolution), and the repertoire of TCR in peripheral blood, HSIL and SCC. Multiplex immunofluorescence technology against distinct immune panels (established within the CTI), will further evaluate the SCC and HSIL immune microenvironments.

The immune-data will be linked to clinical outcome (both radiological and clinical), following radical chemoradiation.

ELIGIBILITY:
Inclusion Criteria:

Males or females, with or without HIV over the age of 18 years at the time of recruitment.

Patients with either:

* A previous complete set of formalin fixed tissue samples of all stages of AIN and anal SCC.
* A new diagnosis of AIN3 and are about to undergo Anal mapping.
* A new diagnosis of Anal Squamous Cell Carcinoma and are about to undergo an Examination under Anaesthetic.

Exclusion Criteria:

* Patients without mental capacity to consent.
* Patients less than 18 years old.
* Patients with anal pathology which is not HPV driven AIN/SCC.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with HPV driven AIN 3 and anal SCC.
Sampling Method: Non-Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2019-04-01 (Actual); Primary Completion 2024-04-30 (Estimated); Study Completion 2024-10-01 (Estimated)

PRIMARY OUTCOMES:
Identify prognostic biomarkers with respect to anal SCC disease progression and treatment response. | 1 year
  Genomic and immune biomarkers
Establish the feasibility of immune analysis and NGS in informing patient treatment decisions. | 1 year
  Pilot study, with low patient numbers

CONTACTS AND LOCATIONS:
Locations (1):
- Imperial College London- Chelsea and Westminster NHS Foundation Trust, London, United Kingdom